CLINICAL TRIAL: NCT03426228
Title: Effects of Fertility Drugs on Glucose Homeostasis and Other Metabolic Parameters on Patients Undergoing In Vitro Fertilization (IVF)
Brief Title: In Vitro Fertilization Impact on Metabolic Parameters
Acronym: IVF
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Collaborators: Fakih IVF Fertility Center (Other); University of Sharjah (Other)
Responsible Party: Principal Investigator, Ayla Coussa, MSc., University of Warwick
Other Study IDs: DSREC-11/2017_09
Record Dates: First submitted 2018-01-03; First posted 2018-02-08 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: GDM; Insulin Resistance; Glucose Intolerance; PCOS; Obesity
Keywords: IVF, Glucose Homeostasis, Metabolic Parameters
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HbA1C — After overnight fasting, 10 ml of blood will be collected at four different timings during the IVF protocol:
  1. At baseline (second day of the menstrual period)
  2. Triggering phase (post-egg retrieval procedure)
  3. Embryo transfer phase (post-transfer procedure)
  4. Week 4 (positive bHCG)
  4. Week 8 of pregnancy
  Other Names: Lipid profile; Hormonal profile: FSH, LH, progesterone, estrogen,Beta-HCG; Serum Insulin level; Fasting Glucose level; Thyroid-Stimulating Hormone

SUMMARY:
A quantitative prospective cohort study will be conducted, where blood samples will be collected at different timings during the IVF protocol, to assess the impact of fertility medications on metabolic parameters of patients undergoing IVF treatment.

DETAILED DESCRIPTION:
Numerous factors predispose women to develop pregnancy-related complications, these include gestational diabetes (GDM), pre-pregnancy obesity, advanced maternal age (> 35 years) and gestational age, abnormal weight gain during pregnancy, family history of diabetes, PCOS and low parity. Evidenced-based studies reported that women with PCOS have a significantly higher risk of developing GDM compared with women without PCOS, independently of the obesity factor; this risk is higher when both factors coexist.

Given the known effect of reproductive hormones on weight-gain, controversies still exist on whether ART predispose women to more adverse obstetric outcomes compared to normal pregnancy. ART describes different procedures to help women become pregnant, with In Vitro Fertilization (IVF) being the most commonly performed. It has been demonstrated that IVF is associated with glucose intolerance in mice and it will be interesting to determine whether this physiologic phenomenon is also altered by IVF medication (such as estrogen and progesterone) in humans. While some studies reported that singleton pregnancies conceived by ART (IVF or ovulation induction) were strongly associated with GDM compared to spontaneous conceptions, other studies did not find significant differences in the risk of GDM. Increased GDM risk presented with IVF can be associated with prenatal obesity or secondary to maternal PCOS condition. The former studies did not specify the body mass index (BMI) and the medical history of participants undergoing IVF, such as the presence of PCOS. Due to limited available data, we still cannot distinguish whether these adverse pregnancy outcomes are due to the pre-existing conditions such as PCOS, or are secondary to the IVF therapy itself.

ELIGIBILITY:
Any patient presenting to us for fresh IVF with the following:

Inclusion Criteria:

* Presenting with or without PCOS
* Presenting with structural or mechanical infertility, such as fallopian tube obstruction, endometriosis, fibroids
* Presenting with male factor
* Presenting with or without insulin resistance
* Combination of more than one of the listed above criteria

Exclusion Criteria:

* Pre-diabetes or diabetes patients (confirmed by impaired or abnormal OGTT)
* Age above 39 years of age
* Taking glucose-lowering meds, such as metformin or janumet.
* Taking corticosteroids

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We will have two main groups of: Obese (BMI: 30-38) and non-obese (BMI: 18.5-29.9) women with the following criteria
Study Population: A convenience sample from adult women of < 39 years of age undergoing fresh IVF treatment at Fakih IVF Clinic in Dubai will be chosen. Participants who will fulfill the inclusion criteria will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Coussa, Dietitian, Principal Investigator — Fakih IVF Dubai
Locations (1):
- Fakih IVF, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
All the study information will be kept confidential. Patients' names will not be identified in any publication or presentation of the study findings. Only groups' results will be reported.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After conducting data collection and analysis the results will be available upon official publication.
Access Criteria: Data access requests will be reviewed by an external independent committee. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Coussa A, Hasan HA, Barber TM. Effects of in vitro fertilization (IVF) therapies on metabolic, endocrine and inflammatory status in IVF-conceived pregnancy. Clin Endocrinol (Oxf). 2020 Dec;93(6):705-712. doi: 10.1111/cen.14270. Epub 2020 Jul 9. PMID 32578220
- [Result] Coussa A, Hasan HA, Barber TM. Impact of contraception and IVF hormones on metabolic, endocrine, and inflammatory status. J Assist Reprod Genet. 2020 Jun;37(6):1267-1272. doi: 10.1007/s10815-020-01756-z. Epub 2020 Mar 25. PMID 32215823

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 702screened -->673eligible to start IVF-->359 had embryo transfer -->191clinically confirmed pregnant+158 negative β-HCG+10 biochem pregnancy--> 64drop-outs+10 miscarriage--> Completed study and included in data: 158 pregnant+117 non-pregnant women
Groups:
- Non-Pregnant: Negative BHCG at 4 weeks
- Pregnant: Positive BHCG at 4 weeks
Period: Overall Study
Arm/Group | Non-Pregnant | Pregnant
Started | 158 | 191
Completed | 117 | 158
Not Completed | 41 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Pregnant | Pregnant | Total
Number analyzed (Participants) | 117 | 158 | 275
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32.5 [25.5 to 39.5] | 32 [25 to 39] | 32.3 [25 to 39.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 158 | 275
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: At 4 weeks, 191 were confirmed pregnant and 158 were non pregnant (negative BHCG). At 12weeks, 117 non-pregnants and 158 pregnants completed the study and analyzed (74 women excluded from data and attributed to drop-outs + those who travelled without completing the 12-week blood test).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 9 | 16 | 25
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 8 | 17
    White | 99 | 134 | 233
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Short-term Effect of Fertility Medications on Glucose Homeostasis and Insulin Resistance in Patients Undergoing IVF Treatment
Description: Participants who experience an abnormal increase in fasting glucose (>110) and A1C (>5.7) will be identified post-treatment. Also, for those previously known to be insulin-resistant, HOMA ratio will help identifying whether the treatment worsens or has no effect on their insulin resistance state.
Time Frame: 12 weeks of pregnancy
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Non-Pregnant | Pregnant
Number analyzed (Participants) | 117 | 158
mg/dL
  Glucose, fasting | 87.62 [79.3 to 95.9] | 82.19 [75 to 89.4]
  Insulin, fasting | 9.37 [4.00 to 14.8] | 9.45 [2.5 to 16.4]

2. Secondary Outcome: Effect of Fertility Medications on Lipids Profile
Description: Lipid profile will be measured before and after treatment; participants experiencing hypercholesterolemia post-treatment will be consulted by a dietitian to help them better manage the condition during their pregnancy (total chol, LDL and triglycerides)
Time Frame: 12 weeks of pregnancy
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Pregnant | Non-pregnant
Number analyzed (Participants) | 158 | 117
mg/dL | 199.5 [155.15 to 243.9] | 174.9 [126.9 to 222.9]

3. Secondary Outcome: Effect of Fertility Medications on Thyroid Function
Description: TSH level will be measured pre- and post-IVF. Early diagnosis of thyroid dysfunction will be closely monitored with frequent repetitions of blood test, especially during the first trimester.
Time Frame: 12 weeks of pregnancy
Measure: Median (Inter-Quartile Range); unit: μIU/mL
Arm/Group | Pregnant | Non-pregnant
Number analyzed (Participants) | 158 | 117
μIU/mL | 1.36 [0.26 to 2.46] | 1.80 [0.75 to 2.85]

4. Other Pre Specified Outcome: Long-term Effect of Fertility Medications in Relation to Maternal and Fetal Outcomes
Description: Early management and/control of metabolic-related adverse outcomes in relation to IVF treatment will prevent GDM by for instance glucophage administration or regular blood test of TSH for participants reported to be at higher risk of thyroid dysfunction.
Time Frame: 9 months of pregnancy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 months
Description: Study is observational and non-experimental. No invasive procedures were used.
Arm/Group | Non-Pregnant | Pregnant
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/158
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/158
Other Adverse Events (participants affected / at risk) | 0/117 | 0/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03426228/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03426228/SAP_001.pdf
  • Informed Consent Form (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT03426228/ICF_002.pdf